CLINICAL TRIAL: NCT01701310
Title: An Open Label Study to Determine the Efficacy of Ferric Carboxymaltose in Preoperative Colorectal Cancer Related Anaemia, and to Develop Biomarkers to Predict Response to This Treatment Strategy
Brief Title: IVICA: Intravenous Iron in Colorectal Cancer Associated Anaemia
Acronym: IVICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11GS005; 2011-002185-21 (EudraCT Number); PB-PG-0110-21041 (Other Grant/Funding Number: RfPB Grant No.)
Record Dates: First submitted 2012-03-21; First posted 2012-10-05 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Anemia; Colorectal Neoplasm
Keywords: Adenocarcinoma; Anemia; Blood Transfusion; Colorectal surgery; Preoperative care; Perioperative care; Postoperative care; Iron; Hematinics; Hepcidin; Quality of life; Postoperative complications
MeSH Terms: conditions — Anemia; Colorectal Neoplasms; Adenocarcinoma; Postoperative Complications | interventions — ferric carboxymaltose; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Experimental)
  Interventions: Drug: Ferric carboxymaltose
- Ferrous Sulphate (Active Comparator)
  Interventions: Drug: Ferrous Sulphate

INTERVENTIONS:
Drug: Ferric carboxymaltose — A minimum of 1 dose of 1000mg of intravenous ferric carboxymaltose will be administered at least 14 days prior to the date of operation.
  Other Names: Ferinject®
  Arms: Ferric carboxymaltose
Drug: Ferrous Sulphate — (Control) 200mg twice a day of oral ferrous sulphate will be administered for a minimum of a two week period
  Arms: Ferrous Sulphate

SUMMARY:
116 eligible patients with confirmed non-metastatic colorectal adenocarcinoma and anemia will be randomized to receive either oral ferrous sulphate (control) or intravenous ferric carboxymaltose (intervention).

It is hypothesized that intravenous iron supplementation is more efficacious than oral iron therapy.

DETAILED DESCRIPTION:
Patients who are anemic at the time of operation have been shown to have an increased frequency of complications including wound infection and longer post-operative admissions. Similarly, patients who are anemic at the time of their cancer operation are more likely to require a blood transfusion which may increase the risk of recurrence of the cancer.

At present, oral iron is often used to treat anemia preoperatively in an attempt to minimize the risk above. This drug is often poorly tolerated due to the side effect profile. Blood transfusions can also be administered but expose the patient to other risks including infection and transfusion associated reactions. In order to overcome these issues, intravenous iron preparations have been developed and have improved in safety.

This is a multi-center, randomized, open label clinical trial, which looks to investigate the efficacy of intravenous iron is in the treatment of preoperative anemia in colorectal patients. Patients will be randomized to receive intravenous ferric carboxymaltose (treatment group) or oral ferrous sulphate (control). The outcomes reviewed will include the amount and frequency of blood transfusions received, changes in patient blood profiles, patient quality of life scores, operative complications and hospital length of stay. The role of hepcidin as a biomarker of treatment response will also be assessed.

The primary hypothesis to be tested is that intravenous iron will decrease transfusion rates. To detect a significant clinical difference in blood transfused consistent with previous published data (1 unit), 58 patients will be required in each arm of the study with 90% power (alpha 0.05).

Randomization will be performed independently to the trial team using a computer generated variable block randomization program.

All data will be confidentially recorded on a Case Report Form, as will drug reactions and side effects.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with histologically proven colorectal adenocarcinoma.
* Anemic at point of diagnosis of colorectal adenocarcinoma. (Haemoglobin values of <12 g/dL for males and <11 g/dL for females)
* Medically fit for surgery.
* Date of planned surgery is >14 days from date of planned initiation of intervention (intravenous ferric carboxymaltose /oral ferrous sulphate).
* Able and willing to comply with all study requirements.
* Willing to allow his/her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion criteria:

* Female participants who are pregnant, lactating or planning a pregnancy during the course of the study.
* Previous gastric, small bowel or colorectal surgery (where ≥50% of stomach or terminal ileum has been resected)
* Current chemotherapeutic treatment.
* Known previous anaemia not attributable to colorectal carcinoma (i.e. anaemia in patients with well established inflammatory disorders or chronic renal disease).
* Known haematological disease.
* Features necessitating urgent surgery (e.g. obstructive symptoms).
* Previous allergy to intravenous iron or related iron products.
* Significant symptomatic anemia necessitating urgent transfusion (e.g. cardiovascular compromise)
* Patients who are unable to consent.
* Significant renal or hepatic impairment.
* -Donation of blood during the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Prisoners and minors (<18 years)
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine if the use of intravenous ferric carboxymaltose can reduce the need for allogeneic blood transfusion compare to oral ferrous sulphate in patients with colorectal adenocarcinoma related anaemia | 0 - 6 to 12 weeks
  To investigate if the number of units transfused per participant, the number of participants whom receive a blood transfusion and the total number of units of blood transfused differs between the two study arms. This period monitored will begin at enrolment into the study, and cease at review in outpatient clinic 6 - 12 weeks post operatively.

SECONDARY OUTCOMES:
To determine differences in hemoglobin and hematinic markers between the groups. | Enrollment to 6-12 weeks postoperatively
  Hematinic markers include ferritin, iron, transferrin, transferrin saturation, erythropoietin.
To determine differences in hepcidin levels in relation to blood profile changes in participants in the intravenous group. | Enrollment to 6-12 weeks postoperatively.
  To review the use of hepcidin as a biomarker to predict response to therapy.
To determine differences in colonic mucosal expression of iron transport proteins, C-myc and NKD1 between the groups | At point of operation only
  Iron transport proteins include DMT TFR1, Ferroportin, Ferritin. As acquired from examination of pathology tissue specimen excised.
To determine differences in postoperative outcomes between the groups. | Enrollment to 6-12 weeks postoperatively
  Post-operative outcomes include morbidity, mortality, length of stay.
To determine differences in anemia symptomatology response between groups. | Enrollment to 6-12 weeks postoperatively
  Quality of Life questionnaires will be used (SF-36[short form 36] and EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Austin G Acheson, MBBS MD FRCS, Study Chair — Nottingham University Hospitals NHS Trust, Nottingham University, School of Clinical Sciences, Division of GI Surgery
Locations (8):
- United Kingdom (8):
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottingham
  - University Hospital Birmingham, Birmingham, West Midlands
  - Royal Wolverhampton Hospitals NHS Trust, Wolverhampton, West Midlands
  - University Hospitals Bristol Foundation NHS Turst, Bristol
  - Derby Hospital NHS Foundation Trust, Derby
  - St James University Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Yeovil District Hospital NHS Foundation Trust, Yeovil